CLINICAL TRIAL: NCT01038323
Title: A Pilot Study on the Combined Use of Cognitive Behavioral Therapy (CBT) and Milnacipran
Brief Title: Drug and Talk Therapy for Fibromyalgia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: IU 0904-08; 1R21AR056046-01A2 (NIH)
Record Dates: First submitted 2009-12-18; First posted 2009-12-23 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; FMS
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CBT and milnacipran (Experimental): Subjects randomized to this group will receive a combination of eight telephone sessions of Cognitive Behavior Therapy (CBT) and a 21-week regimen of milnacipran.
  Interventions: Other: CBT and milnacipran
- CBT and placebo (Placebo Comparator): Subjects randomized to this arm will receive a series of eight telephone sessions of Cognitive Behavioral Therapy (CBT) along with a 21-week regimen of a placebo(sugar pill)medication.
  Interventions: Behavioral: CBT with a placebo
- Educational with milnacipran (Active Comparator): Subjects randomized to this group will receive a series of eight educational phone calls regarding fibromyalgia along with a 21-week regimen of milnacipran.
  Interventions: Drug: Educational with milnacipran

INTERVENTIONS:
Other: CBT and milnacipran — Participants will receive a series of eight telephone sessions of CBT along with a 21-week regimen of milnacipran. Dosing for milnacipran begins with a one week "starter pack". Dosage:12.5 mg on day 1,12.5 mg twice daily on days 2 and 3, then 25 mg twice daily on days 4,5,6,and 7. On day 8 participants will begin taking 50 mg twice daily for the balance of the study.
  Other Names: milnacipran; Savella; Cognitive Behavioral Therapy; CBT; fibromyalgia
  Arms: CBT and milnacipran
Behavioral: CBT with a placebo — Participants will receive a series of eight telephone sessions of CBT along with a 21-week regimen of a placebo. Dosing for the placebo begins with a one week "starter pack". Dosage: 12.5 mg on day 1,12.5 mg twice daily on days 2 and 3, then 25 mg twice daily on days 4,5,6,and 7. On day 8 participants will begin taking 50 mg twice daily for the balance of the study.
  Other Names: placebo; sugar pills; Cognitive Behavioral Therapy; CBT; fibromyalgia
  Arms: CBT and placebo
Drug: Educational with milnacipran — Participants will receive a series of eight telephone sessions of fibromyalgia related education along with a 21-week regimen of milnacipran. Dosing for milnacipran begins with a one week "starter pack". Dosage:12.5 mg on day 1,12.5 mg twice daily on days 2 and 3, then 25 mg twice daily on days 4,5,6,and 7. On day 8 participants will begin taking 50 mg twice daily for the balance of the study.
  Other Names: fibromyalgia; fibromyalgia education; milnacipran; Savella
  Arms: Educational with milnacipran

SUMMARY:
Fibromyalgia Syndrome (FMS) afflicts 2% of the U.S. population and have huge individual and societal costs in terms of quality of life, social and work functioning, health care use, and lost productivity. Although single therapy approaches such as medication, graduated exercise, and Cognitive Behavioral Therapy (CBT) are well-established treatment approaches, the majority of FMS continue to report significant levels of pain and pain-related disability. Testing the efficacy of using combination therapies such and CBT with medication has considerable potential to maximize treatment response. Also, exploring the biological and psychological mechanisms underlying combination treatment may pave the way for developing new treatments for FMS sufferers.

We chose to study drug and CBT for several reasons: 1) the scarcity of trials that manipulate medications along with CBT in FMS, 2) the prohibitive nature of adding an exercise treatment arm in a study that has both time and budgetary constraints, 3) the complexity in understanding the mechanism of actions of 3 different modes of intervention in one clinical trial, and 4) the desire to explore mechanisms in this program of research, in particular the potential effects of a biological intervention (drug) on what is traditionally considered a psychological outcome (pain-related attributions and cognition) and the potential effects of a psychological intervention (CBT) on what is traditionally considered a physiological outcome (pain sensitivity).

DETAILED DESCRIPTION:
Qualified participants will take part in a 21-week clinical research study entitled, "Drug and Talk Therapy for Fibromyalgia". We are doing this study to better understand how talk therapies, such as education and cognitive behavioral therapy (CBT), can improve the therapeutic benefits of drug for fibromyalgia.

Savella ®, (milnacipran) is an FDA approved drug for fibromyalgia. The safety and efficacy of Savella has been established in two US-based clinical studies involving over 2,000 patients with fibromyalgia. Because Savella has already been shown to be effective when used in isolation to treat fibromyalgia, we are conducting the study to determine whether combination treatment (Savella + talk therapy) is more efficacious than just Savella alone or talk therapy alone.

Volunteers will be randomized (like flipping a coin) on two different levels:

1. Each participate will be randomized into one of two groups for medication:

   One group will receive Savella and the other group will receive a placebo (no medicinal value). Both the medication and the placebo will look identical and subjects will not be told into which group they have been placed until the completion of the study. Each participants has 66% chance of receiving Savella and 34% chance of getting the placebo.
2. The second level of randomization will be to determine which type of talk therapies you will be assigned to. Subjects will be randomly assigned to receive educational instruction relevant to fibromyalgia, OR cognitive behavioral therapy which includes a workbook. Both talk therapies will be provided over the phone once a week for 8 weeks. Each phone session may last for 30 minutes. Importantly, both talk therapies can provide coping tools and information designed to help manage fibromyalgia symptoms.

Study Overview:

Subjects will be asked to visit the Fibromyalgia Clinical Research Center on five separate occasions: Initial Screening (today's visit), Week 1, Week 2, Week 9, and Week 21.

VISIT 1:

1. Informed consent and initial screening questionnaire,physical assessment
2. Issue a 'pain score' wrist monitor with instructions to record current pain level three times a day for one week

VISIT 2:

1. Submit your pain recording
2. Complete the self-assessment questionnaires via computer
3. Vital signs check
4. Undergo pain sensitivity testing
5. If qualified, subjects be randomized to receive Savella or placebo AND to receive education or cognitive behavioral therapy

VISIT 3:

1. We will assess the subject's willingness to continue participation.
2. Review medication diary and medication side-effect checklist.
3. Schedule PHONE Therapy sessions: 8 thirty minute calls

VISIT 4:

1. One week prior to this visit, subjects will receive a 'pain score' monitor in order to enter current pain levels three times a day for one week. Then report for this visit.
2. Review side effect checklist, medication diary.
3. Completion of self-assessment questionnaires via computer
4. Undergo pain sensitivity testing

VISIT 5:

1. One week prior to this visit, subjects will receive a 'pain score' monitor in order to enter current pain levels three times a day for one week. Then report for this visit.
2. Review side effect checklist, medication diary.
3. Completion of self-assessment questionnaires via computer
4. Undergo pain sensitivity testing
5. Upon visit completion, participants will receive a reduced dose regimen of the medication along with written and verbal instructions to safely discontinue the study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Must be between the ages of 18 to 65 years of age
2. Must have been diagnosed with fibromyalgia by a rheumatologist
3. Must have an overall body pain average score ≥ 4
4. Must be on stable doses of your current medication for at least past four weeks
5. Must report all medication including herbal supplements and over-the-counter medications that you are currently taking to a member of the research team.
6. Must limit any changes in your medication(s)during the 21-week study time period unless medically necessary
7. Must be willing to maintain a medication diary provided to you during the 21-week study period
8. Must be willing to abstain (not take) any fibromyalgia related medication (including over-the-counter)for at least 6-hours prior to each of the three testing visits. (Otherwise, you may take these medication immediately after pain sensitivity testing has been completed and as prescribed in-between visits)
9. Must experience the symptoms of fibromyalgia syndrome (FMS) that decreases (limits) your ability to perform daily activities.

Exclusions Criteria:

1. You have uncontrolled hypertension(high blood pressure) systolic >160 mm Hg or diastolic blood pressure > 100 mm Hg)
2. If you have a history of: heart disease, glaucoma, or hepatitis
3. You have been diagnosed with any type of peripheral neuropathy
4. You have a body mass index (BMI) of more than 34
5. You currently or frequently have thoughts of harming yourself or committing suicide.
6. You are in the process of filing, or plan to file for disability benefits within the study timeline.
7. You plan to undergo an elective surgery within the study timeline.
8. You have been diagnosed with another major rheumatic conditions (i.e. rheumatoid arthritis, systemic lupus erythematosus, scleroderma and other connective tissue diseases)
9. You are currently pregnant, are planning to become pregnant, or are breastfeeding
10. You have been diagnosed with schizophrenia or manic-depressive.
11. You are currently taking any of the following medications:

    1. fluoxetine, Brand Names: Prozac, Prozac Weekly, Rapiflux, Sarafem
    2. sertraline, Brand Name: Zoloft
    3. paroxetine, Brand Names: Paxil, Paxil CR, Pexeva
    4. citalopram, Brand Name: Celexa
    5. escitalopram, Brand Names: Lexapro
    6. venlafaxine, Brand Names: Effexor, Effexor XR
    7. mirtazapine, Brand Names: Remeron, Remeron SolTab
    8. duloxetine, Brand Name: Cymbalta NOTE: If you are taking any of the medication(s) listed above and are willing to discontinue its use for the duration of this study, you must first discuss your decision with your primary care physician (or prescribing doctor)regarding the appropriate regimen to wean off your current medication and receive his/her written consent before proceeding with enrollment. We will provide you a "Dear Doctor" letter that explains the study details.
12. If you are currently taking or have ever taken Savella® (milnacipran)
13. You are currently participating in other pain research study or have previously been enrolled in any study or class in which cognitive behavioral therapy or educational formats were used to help control pain or stress related to fibromyalgia
14. You are unwilling or unable to comply with the study guidelines

Note: If you have ever experienced an adverse event while taking any type of antidepressant, please alert the research team, while it may not exclude you from participating in the study, it is important that we are aware of the incident in order to keep you safe.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-12; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis C. Ang, MD, Principal Investigator — Indiana University
Locations (1):
- Clinical Research Center for Pain, 250 University Blvd, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] Ang DC, Jensen MP, Steiner JL, Hilligoss J, Gracely RH, Saha C. Combining cognitive-behavioral therapy and milnacipran for fibromyalgia: a feasibility randomized-controlled trial. Clin J Pain. 2013 Sep;29(9):747-54. doi: 10.1097/AJP.0b013e31827a784e. PMID 23446065

RESULTS

PARTICIPANT FLOW:
Groups:
- Combination: Combination cognitive behavioral therapy (CBT) and milnacipran
- Milnacipran: Milnacipran (drug) only
- Cognitive Behavioral Therapy: Cognitive behavioral therapy (CBT) only
Period: Overall Study
Arm/Group | Combination | Milnacipran | Cognitive Behavioral Therapy
Started | 20 | 19 | 19
Completed | 17 | 17 | 15
Not Completed | 3 | 2 | 4
Not completed — Withdrawal by Subject | 3 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination | Milnacipran | Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 20 | 19 | 19 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 19 | 58
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (8.8) | 47.8 (10.6) | 47.11 (11.9) | 46.5 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 16 | 54
  Male | 1 | 0 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 19 | 58
Weekly average pain intensity score [Mean (Standard Deviation); unit: units on a scale] — Average of daily pain scores within a one-week period (scale from 0 to 10, with 10 being the worse possible pain)
  units on a scale | 6.2 (1.2) | 6.3 (1.3) | 6.3 (1.3) | 6.3 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weekly Average Pain Intensity
Description: Change in weekly average pain intensity score from baseline to week 21 (scale from -10 to +10; the more negative the value, the better in terms of pain reduction)
Time Frame: Baseline and Week 21clinic visits
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Combination | Milnacipran | Cognitive Behavioral Therapy
Number analyzed (Participants) | 17 | 17 | 15
units on a scale | -2.1 (.43) | -0.97 (0.43) | -1.67 (0.45)

2. Secondary Outcome: Change in Evoked Pain Scores
Description: 0 to 20 pain scale, with higher pain score representing greater sensitivity to pressure pain stimuli
Time Frame: Baseline and Week 21 clinic visits
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Combination | Milnacipran | Cognitive Behavioral Therapy
Number analyzed (Participants) | 17 | 17 | 15
units on a scale | -0.76 (1.2) | -0.41 (1.2) | 0.78 (1.2)

3. Secondary Outcome: Identification of Group Assignment
Description: Subjects identifying group assignment correctly
Time Frame: week 21
Population: Information not captured (unfortunately)
Measure: Number; unit: participants
Arm/Group | Combination | Milnacipran | Cognitive Behavioral Therapy
Number analyzed (Participants) | 17 | 17 | 15
participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 21 weeks
Groups:
- Combination: Cognitive behavioral therapy + milnacipran
- Milnacipran: milnacipran + education
- Cognitive Behavioral Therapy: Cognitive behavioral therapy + placebo
Arm/Group | Combination | Milnacipran | Cognitive Behavioral Therapy
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 9/20 | 8/19 | 3/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination (N=20) | Milnacipran (N=19) | Cognitive Behavioral Therapy (N=19)
nausea (Gastrointestinal disorders) | 9 (9) | 8 (8) | 3 (3) — transient nausea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No